CLINICAL TRIAL: NCT00006218
Title: A Phase I Study of 3-Aminopyridine-2-Carboxaldehyde Thiosemicarbazone (3-AP, Triapine) in Cancer Patients Using a 96-Hour Intravenous Continuous Infusion
Brief Title: 3-AP in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vion Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: VION-CLI-009; CDR0000068067 (Registry Identifier: PDQ (Physician Data Query)); AECM-12000041110; NCI-V00-1598
Record Dates: First submitted 2000-09-11; First posted 2004-03-17 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2007-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — 3-aminopyridine-2-carboxaldehyde thiosemicarbazone

INTERVENTIONS:
Drug: triapine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of 3-AP in treating patients who have advanced cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety, tolerability, and toxicity of 3-AP in patients with advanced malignancies. II. Determine the maximum tolerated dose and recommended phase II dose of this treatment in these patients. III. Determine the pharmacokinetic parameters of this treatment in these patients. IV. Determine the tumor response in these patients treated with this regimen.

OUTLINE: This is a dose escalation, multicenter study. Patients receive 3-AP IV continuously over 96 hours. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients with complete response receive treatment for 1 course past the course in which the complete response was documented; patients with partial response may receive treatment for up to 1 year; and patients with stable disease may receive treatment for up to 6 months. During the accelerated phase of the study, cohorts of 1 patient each receive escalating doses of 3-AP until one patient experiences dose limiting toxicity (DLT) or 2 different patients experience grade 2 toxicity during any course. When the accelerated phase ends, cohorts of 3-6 patients receive escalating doses of 3-AP until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience DLT.

PROJECTED ACCRUAL: Approximately 21 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced or metastatic malignancy Failed one or more prior standard therapies or considered unlikely to respond to any currently available therapy Measurable or evaluable disease No active, untreated CNS metastases (stable for at least 2 months and no evidence of new CNS metastases)

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: Greater than 3 months Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 10 g/dL (transfusion allowed) No bleeding disorder (except occult blood for gastrointestinal cancers) Hepatic: Bilirubin no greater than 2.0 mg/dL ALT, AST, and alkaline phosphatase no greater than 3 times upper limit of normal (ULN) (no greater than 5 times ULN with liver metastases) PT and PTT no greater than 1.5 times ULN Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No active heart disease No myocardial infarction within the past 3 months No symptomatic coronary artery disease or heart block No uncontrolled congestive heart failure Pulmonary: No moderate to severe compromise of pulmonary function Other: No active infection No mental deficits and/or psychiatric history that would preclude study No other concurrent life threatening illness Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 18 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered No persistent chronic toxicity from prior chemotherapy greater than grade 1 Endocrine therapy: Not specified Radiotherapy: At least 3 weeks since prior radiotherapy Concurrent radiotherapy to single site of progressive disease allowed during first course of study treatment Surgery: Not specified Other: At least 3 weeks since any prior treatment for malignancy and recovered No other concurrent investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-05; Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Sznol, MD, Study Chair — Vion Pharmaceuticals
Locations (1):
- Albert Einstein Comprehensive Cancer Center, The Bronx, New York, United States